CLINICAL TRIAL: NCT00815009
Title: Prospective Histopathologic Evaluation of Diet and Exercise in Patients With Non-Alcoholic Fatty Liver Disease
Brief Title: Evaluation of Diet and Exercise in Patients With Non-Alcoholic Fatty Liver Disease
Acronym: NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Renee E. Cole, Director, US Military Dietetic Internship Consortium, San Antonio Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2008.171
Record Dates: First submitted 2008-12-24; First posted 2008-12-29 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Fatty Liver
Keywords: NAFLD; NASH
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Std of Care) (No Intervention): Standard of Care/Control, including Lifestyle Advice (attend a basic healthy nutrition class as well as follow up appointments with GI MD).
  Interventions: Behavioral: Mod Fat/Low Processed Carb Diet and Moderate Exercise
- B (Low Fat) (Experimental): Standard of Care, plus Low Fat Diet and Moderate Exercise
  Interventions: Behavioral: Mod Fat/Low Processed Carb Diet and Moderate Exercise; Behavioral: Low Fat Diet and Moderate Exercise
- C (Mod Fat) (Experimental): Standard of Care, plus Moderate Fat/Low Processed Carbohydrate Diet and Moderate Exercise
  Interventions: Behavioral: Mod Fat/Low Processed Carb Diet and Moderate Exercise
- D (Exercise only) (Experimental): Standard of Care plus Moderate Exercise only
  Interventions: Behavioral: Mod Fat/Low Processed Carb Diet and Moderate Exercise; Behavioral: Moderate Exercise Only

INTERVENTIONS:
Behavioral: Mod Fat/Low Processed Carb Diet and Moderate Exercise — Follow a moderate fat with low processed carbohydrate diet with moderate exercise at the cardiac rehab clinic (2x/wk for 8 wks, 1x/wk for 8 wks, 1x/2wks for 8 wks)
  Other Names: Low Carb / Mod Fat
Behavioral: Low Fat Diet and Moderate Exercise — Follow a low fat diet along with moderate exercise at the cardiac rehab clinic (2x/wk for 8 wks, 1x/wk for 8 wks, 1x/2wks for 8 wks)
  Other Names: Low Fat
  Arms: B (Low Fat)
Behavioral: Moderate Exercise Only — No special dietary meal plan. Moderate exercise in the cardiac rehab clinic (2x/wk for 8 wks, 1x/wk for 8 wks, 1x/2wks for 8 wks)
  Other Names: Mod exercise
  Arms: D (Exercise only)

SUMMARY:
Moderate exercise with a low fat and/or a moderate fat with low processed carbohydrate diet will have a greater effect on slowing disease progression and reversing hepatic steatosis and/or necro-inflammation in the liver of adult patients with NAFLD and NASH when compared to a regular healthy diet alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* DEERS eligible (DoD beneficiary)
* All participants must plan to be in the area for at least nine months
* Liver biopsy confirmed NAFLD/NASH (NAS Score evaluating steatosis, lobular inflammation and hepatocyte ballooning) within the past 6 months

Exclusion Criteria:

* Alcohol consumption > 20 g/d or history of alcohol abuse
* Hepatitis A, B, C
* Chronic liver disease of any other etiology
* Fatty acid oxidation disorder (Inborn errors of metabolism)
* Insulin therapy regime for treatment of diabetes
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
NAFLD Activity Score (Percent liver steatosis, inflammation, and fibrosis) | 6 months

SECONDARY OUTCOMES:
Insulin resistance (IR) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Renee E Cole, MS, PhD, Principal Investigator — San Antonio Military Medical Center
Locations (1):
- San Antonio Military Medical Center, Fort Sam Houston, Texas, United States